CLINICAL TRIAL: NCT05987891
Title: The Influence of Cardiovascular Risk Factors on Electrocardiographically and Hemodynamics Responses to Treadmill Exercise Test in Asymptomatically Subjects: a Clinical Perspective (ERGO-RISC)
Brief Title: Cardiovascular Risk Factors on Electrocardiographically and Hemodynamics Responses to Treadmill Exercise Test
Acronym: ERGO-RISC
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Pedro Gabriel Senger Braga, Ph.D., University of Sao Paulo
Other Study IDs: Pró-Coração
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Abnormalities; Healthy
Keywords: treadmill exercise test; asymptomatic subjects; Cardiovascular risk factor
MeSH Terms: conditions — Cardiovascular Diseases; Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy controls: Volunteers will perform treadmill exercise tests. It will be monitored electrocardiogram, heart rate, and blood pressure in the rest state, under exercise, and in the recovery.
  Interventions: Diagnostic Test: Treadmill exercise stress test

INTERVENTIONS:
Diagnostic Test: Treadmill exercise stress test — Ellestad protocol will be applied in all subjects up to fatigue and recovery will be monitored.

SUMMARY:
The goal of this observational cross-sectional study is to analyze the effect of cardiovascular risk factors in healthy and asymptomatic populations. The main questions it aims to answer are:

* Does the combination of the presence of different risk factors increase the risk for abnormalities appearing on electrocardiograms, such as ischemia, arrhythmia, and hemodynamics effects during and at the peak of effort of treadmill exercise test?
* What are the main differences observed in the recovery period? Participants will answer an anamnesis of risk factors such as sex, race, age, familiar history of coronary artery disease, overweight or obesity, smoking, stress, and physical activity practice and perform treadmill exercise test on Ellestad protocol. If there a comparison groups: Researchers will compare individuals with most risk factors with those without, to see the cardiovascular responses.

DETAILED DESCRIPTION:
The main outcomes broad the effect of simples and easy doccumented cardiovascular risk factors such as sex, race, age, familiar history of coronary artery disease, overweight or obesity, smoking, stress, and physical inactivity on electrocardiogram and hemodinamics abnormalities during and after exercise treadmill exercise test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that can complete the treadmill exercise test with the Ellestad protocol with 6 minutes of recovery.

Exclusion Criteria:

* Use of remedies for blood pressure, glycemia, cholesterol, and serum lipids;
* Symptomatically subjects;
* Electrocardiogram that are not able to be interpreted;
* Blood pressure in rest state ≥180 mmHg and ≥110 mmHg, for systolic and diastolic, respectively.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy and assymptomatically subjects who are visiting cardiologyst for routine.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
ECG abnormalities and risk factors | 1 year
  Electrocardiogram suggestive of myocardial ischemia

CONTACTS AND LOCATIONS:
Locations (1):
- Pró-Coração, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Almeida Dourado JP, Azevedo LM, de Almeida Dourado L, de Oliveira JG, de Faria BB, de Oliveira Matos K, Roever L, Dourado PMM, Braga PGS. Association Between Psychosocial Stress and Premature Ventricular Contractions During the Recovery Phase Following Treadmill Testing in Asymptomatic Individuals. J Clin Med. 2025 Jun 30;14(13):4637. doi: 10.3390/jcm14134637. PMID 40649011